CLINICAL TRIAL: NCT00794560
Title: Self-management of Heparin Therapy - Drug Use Problems and Compliance With Self-injected Low Molecular Weight Heparin in Ambulatory Care
Brief Title: Self-management of Low Molecular Weight Heparin Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NRA 630 00 23; EKBB 95/07 (Other: ethics committee)
Record Dates: First submitted 2008-11-18; First posted 2008-11-20 (Estimated); Results first posted 2014-08-13 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Thromboembolism
Keywords: Heparin, Low-Molecular-Weight; compliance; drug safety; self-administration; ambulatory Care; Pharmaceutical Services
MeSH Terms: conditions — Thromboembolism; Patient Compliance | interventions — Patient Education as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- clinical setting: intervention (Experimental): Recruitment of patients in the hospital into the randomized intervention group. Intervention is done by a trained pharmacist/Doctor of Philosophy-student in the study center (a pharmacy) or at patient's bedside in the hospital.
  Intervention: patient education
  Interventions: Behavioral: patient education
- clinical setting: standard care (No Intervention): Recruitment of patients in the hospital into the randomized control group (standard care in community pharmacy)
- daily life setting: intervention (Experimental): Recruitment of patients in trained community pharmacies into the intervention group. Intervention is done by trained pharmacists.
  Intervention: patient education
  Interventions: Behavioral: patient education
- daily life setting: standard care (No Intervention): Recruitment of patients in community pharmacies into control group (standard care in community pharmacy)

INTERVENTIONS:
Behavioral: patient education — Possible, individualized interventions:
  * Improvement of patient's knowledge about medication, therapy and drug application by providing detailed written information material
  * Providing a complete equipment package for self-injection (disinfection patches, patches, plasters, waste disposal box for used syringes)
  * Patient training: oral instructions for self-injection (and application, if required), exercising the injection technique on a phantom
  * First self-injection under control of a specially trained pharmacist
  Arms: clinical setting: intervention; daily life setting: intervention

SUMMARY:
There is very little data available on compliance with self-injected low molecular weight heparins (LMWH), but what there is, definitely shows that compliance represents a significant problem. We therefore aim to a) record drug use problems of patients including compliance, b) develop a "SOP" for first instruction by a pharmacist and for subsequent pharmaceutical care and c) to compare intensive pharmaceutical care (intervention) vs. standard care (control) provided in the pharmacy to patients with a prescription for a LMWH as an outpatient treatment.

Hypothesis:

Intensive pharmaceutical care in ambulatory patients who self-inject low molecular weight heparins results in improved compliance, more safety and satisfaction as well as in fewer complications.

DETAILED DESCRIPTION:
Patient recruitment in community pharmacies enables the testing of the feasibility of the interventions under daily-practice conditions and facilitates the recruitment of a larger number of patients.

Data collection:

* telephone interviews with structured questionnaires at the beginning and at the end of the therapy
* monitored self-injection in the study center or at patient's home (direct observation technique [DOT])
* compliance measurement: answers from patient interviews, comparing number of used syringes vs. number of prescribed syringes (analogue "pill count"), measuring residual volume in recycled syringes
* recording of the fine motor skills by the adapted "Disabilities of the Arm, Shoulder and Hand" questionnaire (DASH questionnaire)

ELIGIBILITY:
Inclusion Criteria:

* Patients are recruited from orthopedic clinics, an emergency department and from community pharmacies with a prescription for a LMWH as an outpatient treatment.
* self-application of the LMWH
* german / english speaking

  -> clinical setting:
* Dalteparin

  -> daily life setting:
* all LMWH (ready-to-use syringes)
* control group: self-application or application by another person (family member, medical person, etc.)

Exclusion Criteria:

- patient's home far away from study center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2007-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kurt E. Hersberger, Prof. PhD, Principal Investigator — Pharmaceutical Care Research Group, University of Basle, Switzerland
Locations (2):
- Switzerland (2):
  - University Hospital of Basle, Switzerland, Basel
  - Kantonsspital Baselland, Switzerland, Bruderholz

REFERENCES:
- [Result] Mengiardi S, Tsakiris DA, Molnar V, et al. Impact of Pharmaceutical Care on Self-Administration of Outpatient Low-Molecular-Weight Heparin Therapy. Pharmacology & Pharmacy 5: 372-385, 2014

RESULTS

PARTICIPANT FLOW:
Groups:
- Clinical Setting: Intervention: Recruitment of patients in the hospital into the randomized intervention group. Intervention is done by a trained pharmacist/Doctor of Philosophy-student in the study center (a pharmacy) or at patient's bedside in the hospital.
  patient education: Possible, individualized interventions:
  * Improvement of patient's knowledge about medication, therapy and drug application by providing detailed written information material
  * Providing a complete equipment package for self-injection (disinfection patches, patches, plasters, waste disposal box for used syringes)
  * Patient training: oral instructions for self-injection (and application, if required), exercising the injection technique on a phantom
  * First self-injection under control of a specially trained pharmacist
- Daily Life Setting: Intervention: Recruitment of patients in trained community pharmacies into the intervention group. Intervention is done by trained pharmacists.
  patient education: Possible, individualized interventions:
  * Improvement of patient's knowledge about medication, therapy and drug application by providing detailed written information material
  * Providing a complete equipment package for self-injection (disinfection patches, patches, plasters, waste disposal box for used syringes)
  * Patient training: oral instructions for self-injection (and application, if required), exercising the injection technique on a phantom
  * First self-injection under control of a specially trained pharmacist
Period: Overall Study
Arm/Group | Clinical Setting: Intervention | Clinical Setting: Standard Care | Daily Life Setting: Intervention | Daily Life Setting: Standard Care
Started | 36 | 36 | 44 | 38
Completed | 33 | 32 | 40 | 34
Not Completed | 3 | 4 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clinical Setting: Intervention | Clinical Setting: Standard Care | Daily Life Setting: Intervention | Daily Life Setting: Standard Care | Total
Number analyzed (Participants) | 33 | 32 | 40 | 34 | 139
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 56 [34 to 60] | 56 [42 to 66] | 51 [36 to 65] | 54 [43 to 67] | 54 [40 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 17 | 18 | 70
  Male | 17 | 13 | 23 | 16 | 69

OUTCOME MEASURES:

1. Primary Outcome: Drug Use Problems
Description: During a home visit and at her/his individual injection time, each patient was monitored when self-administering an s.c. injection (directly observed therapy, DOT). Score minimum = -2.00; score maximum = +2.00 for the objective estimation of the application quality. Higher score values represent better outcomes.
Time Frame: during the individual drug therapy, an average of 18 days
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Clinical Setting: Intervention | Clinical Setting: Standard Care | Daily Life Setting: Intervention | Daily Life Setting: Standard Care
Number analyzed (Participants) | 33 | 32 | 40 | 34
scores on a scale | 1.25 (0.27) | 0.86 (0.33) | 1.20 (0.41) | 1.17 (0.40)

2. Secondary Outcome: Compliance
Description: objectively determined by syringe count Therapy durations varied individually depending on the indication of the drug therapy (days to weeks).
Time Frame: at the end of the individual drug therapy, an average of 18 days
Measure: Mean (Standard Deviation); unit: percentage of syringes
Arm/Group | Clinical Setting: Intervention | Clinical Setting: Standard Care | Daily Life Setting: Intervention | Daily Life Setting: Standard Care
Number analyzed (Participants) | 33 | 32 | 40 | 34
percentage of syringes | 94.5 (10.5) | 96.2 (10.6) | 95.1 (10.0) | 97.5 (4.2)

3. Secondary Outcome: Patient Satisfaction
Time Frame: at the end of the individual drug therapy, an average of 18 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: During the entire individual s.c. injection therapy, up to 6 weeks.
Description: Therapy durations varied individually depending on the indication of the drug therapy (days to weeks).
Arm/Group | Clinical Setting: Intervention | Clinical Setting: Standard Care | Daily Life Setting: Intervention | Daily Life Setting: Standard Care
Serious Adverse Events (participants affected / at risk) | 0/36 | 1/36 | 0/44 | 0/38
Other Adverse Events (participants affected / at risk) | 33/36 | 29/36 | 37/44 | 17/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clinical Setting: Intervention (N=36) | Clinical Setting: Standard Care (N=36) | Daily Life Setting: Intervention (N=44) | Daily Life Setting: Standard Care (N=38)
Allergy / hypersensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — hospitalisation due to allergy, completely recovered
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clinical Setting: Intervention (N=36) | Clinical Setting: Standard Care (N=36) | Daily Life Setting: Intervention (N=44) | Daily Life Setting: Standard Care (N=38)
hematoma at injection site (Skin and subcutaneous tissue disorders) | 31 (31) | 26 (26) | 35 (35) | 15 (15)
mild injection site irritation/burning (Skin and subcutaneous tissue disorders) | 16 (16) | 17 (17) | 22 (22) | 5 (5)
hematoma in general (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 5 (5) | 3 (3)
site pain (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 4 (4) | 3 (3)
induration (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0) | 3 (3) | 0 (0)
exanthema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No